CLINICAL TRIAL: NCT02662426
Title: Randomized, Double-Blinded, Oseltamivir-and-Placebo-Controlled Clinical Study About Lingdancao Granules in the Treatment of Seasonal Influenza
Brief Title: Lingdancao Granules in the Treatment of Seasonal Influenza
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Hongxia Ma, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IFLDCRct
Record Dates: First submitted 2015-11-01; First posted 2016-01-25 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Influenza
Keywords: Seasonal Influenza; Lingdancao; RCT
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Drugs for experimental group (Experimental): Lingdancao granules, 4 packs per time (3g/pack), three times per day; analogous oseltamivir phosphate capsule, 1 capsule per time, twice per day.Drugs must be used on the day of fever and last for five days continuously.
  Interventions: Drug: Lingdancao granules; Drug: analogous oseltamivir phosphate capsule
- Drugs for positive control group (Active Comparator): Oseltamivir phosphate capsule (tamiflu), 1 capsule per time (75mg), twice per day; analogous Lingdancao granules, 4 packs per time, three times per day.Drugs must be used on the day of fever and last for five days continuously.
  Interventions: Drug: Oseltamivir phosphate capsule; Drug: analogous Lingdancao granules
- Drugs for placebo control group (Placebo Comparator): Analogous Lingdancao granules, 4 packs per time, three times per day, analogous oseltamivir phosphate capsule, 1 capsule per time, twice per day.Drugs must be used on the day of fever and last for five days continuously.
  Interventions: Drug: analogous oseltamivir phosphate capsule; Drug: analogous Lingdancao granules

INTERVENTIONS:
Drug: Lingdancao granules — 4 packs per time (3g/pack), three times per day
  Other Names: Lingdancao granules,z53021634
  Arms: Drugs for experimental group
Drug: analogous oseltamivir phosphate capsule — 1 capsule per time, twice per day
  Other Names: analogous oseltamivir phosphate capsule,0221503013
  Arms: Drugs for experimental group; Drugs for placebo control group
Drug: Oseltamivir phosphate capsule — 1 capsule per time (75mg), twice per day
  Other Names: tamiflu,0221503013
  Arms: Drugs for positive control group
Drug: analogous Lingdancao granules — 4 packs per time, three times per day
  Other Names: analogous Lingdancao granules,z53021634
  Arms: Drugs for placebo control group; Drugs for positive control group

SUMMARY:
Name of study:

Randomized, Double-Blinded, Oseltamivir-and-Placebo-Controlled Clinical Study about Lingdancao Granules in the Treatment of Seasonal Influenza

Objective:

Preliminary evaluation on the efficacy and safety of Lingdancao granules in the treatment of seasonal influenza

Design:

Multicenter, randomized, double-blind, double parallel analogy, positive drug and placebo controlled trial

Case number:

This test is expected to be included in 318 cases of 14-65 (≥14 or ≤65) ages of subjects. Qualified participants are randomly divided into experimental drug group (Lingdancao granules group), positive control group (oseltamivir phosphate group) and placebo group, 106 cases in each.

DETAILED DESCRIPTION:
Study Objectives This study wishes to evaluate the efficacy and safety of Lingdancao granules for the treatment of seasonal influenza (including seasonal influenza A/H1N1 and A/H3N2 type, the new influenza A (H1N1) or influenza B) and an economic analysis on drugs in an evidence-based clinical trial with Oseltamivir phosphate Capsules and placebo as contrast.

Design and Trial registration This clinical study is a multicentered, randomized, double-blind, double control trial that testes drugs and placebo. Non-inferiority (vs. positive control) and superiority (vs. placebo control) trials are conducted.

After clinical ethics approval and before the participants' randomly enrolment, the research plan is registered both in clinicaltrials.gov and in the center of Chinese clinical trial.

Study participants

1 Designed case number of participants The study is designed to enroll 360 411 cases of patients (male and female) suffering seasonal influenza (including seasonal influenza type A/H1N1 and A/H3N2, the new influenza A (H1N1) or influenza B) aged 14-65 years.

Recommendations from the World Health Organization (WHO) for influenza-like illnesses (ILIs) are used as the basis for influenza surveillance. If a patient presents with an acute cough and fever, clinicians must be highly vigilant to test for infections caused by the influenza virus. In general, the rate of ILI cases that lead to a clinical diagnosis of influenza infection is about 18-80%, which is higher than other clinical diagnoses, e.g. acute infections of the upper respiratory tract. Therefore adult ILI patients are selected for inclusion in the study.

Treatment

1. Drugs 1.1 Drugs for experimental group Lingdancao granules (3g/pack, license number XXXXX, produced by Panlongyunhai Co., Ltd.) 1.2 Drugs for control group Oseltamivir phosphate capsule (tamiflu) (License number J20090076, produced by Shanghai Lou's Pharmaceutical Co., Ltd.) 1.3 Analogous drugs Analogous Lingdancao granules (license number XXXX) Analogous oseltamivir phosphate capsule (license number XXXX) All drugs are packaged by the Panlongyunhai Co., Ltd. according to the requirements of a double-blind, double-simulation test.
2. Dosage and specifications 2.1 Study drugs Lingdancao granules, electuary (IIR, 3g/pack, license number XXXXX, produced by Panlongyunhai Co., Ltd.) Oseltamivir phosphate capsule (tamiflu) (98.5mg/capsule, equals to 75mg oseltamivir, license number J20090076) Placebo, analogous Lingdancao granules, analogous oseltamivir phosphate capsule (specifications as above, produced by Panlongyunhai Co., Ltd.) Randomly numbered ①②③, prescribed by doctors according to the selected time sequence of the patients 2.2 Package and label All drugs are packaged by the Panlongyunhai Co., Ltd. according to the requirements of a double-blind, double-simulation test, in order to avoid patients to differentiate the three. All drugs will be packed by randomly number①②③ with 5 days dosage. Each pack has 2 parts of viscous labels, including parts for peeling off. Drug labels will be printed in Chinese, including following contents.

   * Study plan registration number
   * Random number/drug number
   * Subject initials
   * Drug specifications
   * Usage and dosage (medication guidance)
   * Storage conditions (storage temperature)
   * Avoid children taking by mistake
   * Date of dispensing
   * Only for use of clinical research
   * Name of bidding company 2.3 Random blind coding and distribution Participants will be randomly assigned into the experimental group or control group in accordance with sequence of selecting. Random Numbers must be in sequence from small to large, with no missing or wrong number, otherwise will be in violation of the design.

   2.4 Blinded study and evaluating time This study is a randomized blinded parallel controlled clinical trial, designed by statistical professionals using computer simulation for random scheme. The preparation of blind coding and treatment code is completed according to regulations, and corresponding report of blind coding record is completed and preserved in duplicate, respectively at the sponsor and clinical trials group units.

   Subjects through screening are entered into the stage of blinded study when drugs are dispending according to the random number sequence by a researcher at the specified, Researchers participating in symptom evaluation have no knowledge of the kind of study drugs.
3. Usage and dosage Dosing based on instructions of Lingdancao particles and Oseltamivir phosphate capsules (tamiflu).

3.1 Drugs for experimental group Lingdancao granules, 34 packs per time (3g/pack), three times per day; analogous oseltamivir phosphate capsule, 1 capsule per time, twice per day 3.2 Drugs for positive control group Oseltamivir phosphate capsule (tamiflu), 1 capsule per time (75mg), twice per day; analogous Lingdancao granules, 34 packs per time, three times per day 3.3 Drugs for placebo control group Analogous Lingdancao granules, 4 packs per time, three times per day Analogous Lingdancao granules, 3 packs per time, three times per day, analogous oseltamivir phosphate capsule, 1 capsule per time, twice per day 4 Course of treatment Drugs must be used on the day of fever and last for five days continuously. In addition, in view of the contagiousness of virus, take 2 days after prior symptoms disappear as the boundary, is possible to continue medical treatment after the participants' symptoms disappear.

Participators who meet the inclusion criteria are given by the study drugs according to the random number on the day when they are included into the study. And the first day using drugs is defined as the first day of the study, while the second day begins from 24:00 the same day. According to the time of the first medication, the last time for using drug will be on the 5th or 6th day. If the first medication is after 17:00 on the first day, the next meditation will be on the following morning. In this case, the last medication will be on the morning of the 6th day. If the first medication is before 17:00 on the first day, the next administration will be on the same day at night (before midnight). In this case, the last time to give medicine will be in the evening on the 5th day.

5 Other treatment Once other drugs are taken because of inevitable condition, or dosage is changed, the name of drug, reason for using, methods, dose and time of using must recorded on the case table.

5.1 Standard of drug using Body temperature≥38.5℃, cannot be lower after 4 hours' physical cooling, or body temperature gradually raised up to more than 39℃; or headache, muscle pain symptom scores 3 points or more.

5.2 Symptomatic drugs (provided by the Panlongyunhai Company) 5.2.1 Fever, acetaminophen. 5.2.2 Cough with white phlegm, brombexine hydrochloride. 5.2.3 Mild asthma, long-term theophylline. Apart from the drug above, no other drugs can be used. 6 Criteria for free additional auxiliary examination 6.1 In case of worsening cough, phlegm, bloody sputum, chest pain or fast breathing rate, dyspnea, routine blood test, chest X-ray examination are given; 6.2 In case of gastrointestinal symptoms such as vomiting, diarrhea, routine blood test, liver function, renal function, blood electrolyte are given; 6.3 In case of heart palpitation, chest suppression, chest pain and syncope, electrocardiogram (ECG) and myocardial enzyme are given.

7 Compliance Researchers or co-researchers will guide participants record the actual dose of drugs in their diary. According to the diary, researchers or co-researchers will evaluate compliance of the participant on the basis of the following four grades in different stages and record it in the case report after each follow-up.

7.1 Take medications according to rules. 7.2 Take medications mostly according to rules, (80%-120% of the designed dose) 7.3 Take medications half of the time according to rules. 7.4 Almost with no medication (no more than half the time) Once the subject is not taking drugs according to stipulations, reasons must be indicated.

Because of the particularity of influenza, doctors can keep the subjects hospitalized until the fever is retreated according to specific conditions.

Study design 1 General design and arrangement This study will follow design of randomized, blinded, positive drug and placebo controlled together with parallel group; subjects are screened from seasonal influenza virus infected patients.

300 411patients conforms to the inclusion and exclusion criteria and signed informed consent are participating in this study, and are randomly assigned to Lingdancao granules group, Oseltamivir phosphate capsules (Tamiflu) group, and placebo group.

2 Specific processes Follow-up Visit 1 0 Screening and baseline Before the start of the trial, patients should be fully obtain written and verbal descriptions about the study, and signed a written informed consent.

Record

1. Demographic information

   - History (history of influenza, exposure history, history of other diseases treatment)
2. - Physical examination

   * Evaluation of flu-like symptoms
   * Temperature measurement
   * Regular blood pressure and pulse measurement
3. - Laboratory tests

   * Routine blood test, liver function test of three, renal function test of two, blood electrolytes, myocardial enzyme, blood sugar tests
   * Virus nucleic acid, separation, virus antigen and serologic test
   * Women of childbearing age with pregnancy test (urine pregnancy test)
   * 12 - lead electrocardiogram (ECG)
4. - Distribution of diary
5. - Record of any other drugs along the course Patients meeting the inclusion criteria will be distributed of 1 week medication of blinded study, and be recorded in the release/return registration form. These patients will be randomly assigned into the three 3 treatment groups (Lingdancao group , Tamiflu group and placebo group), with random number provided by West China Hospital of Sichuan University Evidence-based Medicine Centers. Subjects are informed to take the medication according to a corresponding method from the day on. All patients attending the screening shall be recorded on the including table. Reasons for not included should be recorded.

Laboratory tests given before follow-up1 up0 are used for screening subjects into the research, as well as a baseline of other laboratory tests.

Follow-ups 21-5 3 are treatment period. Each of the follow-up should include the following.

* Evaluation of the degree of influenza-like symptoms, the time required and time for defervescense of the patients from their diary
* Record of the drug distribution and the number of returned pills on the drug issue/return registration form, and evaluate the compliance. Once there's quantity discrepancy, reasons need to be recorded.
* Record of other drugs along the treatment
* Record of any adverse events
* Instruction of subjects' medication according to the study process. In case of twice of adverse events occurrence between two follow-ups, researchers should be informed as soon as possible.
* Instruction of bringing back the drug box at each follow-up for compliance evaluation. If drug dose adjustment happened between two follow-ups, the factors should be considered in the compliance evaluation.

Follow-up7 up 4 or premature termination need to carriy out the following.

* Evaluation of influenza-like symptoms
* Temperature measurement
* Record of the drug distribution and the number of returned pills on the drug issue/return registration form, and evaluate the compliance. Once there's quantity discrepancy, reasons need to be recorded.
* Record of other drugs along the treatment
* Record of any adverse events
* Physical check
* Regular blood pressure and pulse measurement
* 12- lead electrocardiogram (ECG)
* Laboratory tests Routine blood test, liver function of three, renal function of two, blood electrolytes, myocardial enzyme, blood sugar test Virus nucleic acid, separation test Serologic test
* Conclusions of the subject's treatment
* Overall evaluation of clinical curative effect 3 Study Scheme 3.1 Visit plan On the 3rd, 5th, 7th and 21st days after the first visit patients shall have follow-ups in person while the rest by telephone. The time windows of follow-up 3rd, 5th, 7th days are +1 day, and for 21st day is +7 days.

Study medications, other drugs and basic treatment should be given by the doctors or taken according to the doctor's guidance; participants will receive a written guidance about the daily usage of the drugs.

Participants should report daily to researchers about the number of pills taken. In addition, the researchers need to count the number of pills in the opened drug boxes, and the number of unpacking boxes. After the test, all the rest of the study drug or placebo must be returned to the clinical arbitrator together with boxes.

3.2 Principles and standards of suspending After starting taking study drug, once any of the following circumstances appear, the researchers or co-researchers must stop the treatment of patients and take corresponding measures immediately.

* Symptom aggravating and cannot continue taking the drugs (diagnosis and treatment refer to Diagnosis and Treatment of Influenza Manual (2011 edition))
* Adverse events that cannot continue taking the drugs (including abnormal blood pressure, pulse, laboratory values, and ECG with clinical significance)
* Other conditions that researchers or co-researchers think should terminate the treatment Cause of suspending the study in advance should be recorded. Subjects suspended from the study must complete all contents of follow-up7 (or ending examinations and tests).

3.3 Shedding and missing follow-ups After the beginning of the study's medication, once the subjects drop out the study due to any of the following reasons, the researchers or co-researchers must take the appropriate measures and investigate the result of the subjects.

* Participants wish to quit the study
* During the study, subjects stop the follow-up to the hospital for none-direct related reasons, such as transferring to another hospital or address migration.

3.4 Principles and standards for comprehensive stopping of the study

1. Serious security problems in the study
2. Study finds that the drugs' effect are so poor or even invalid, that should suspend the study.
3. Significant errors or important deviation appears in the clinical trial scheme, and it's difficult to evaluate effect of the drugs.
4. The sponsor required for an end (due to reasons of funds, management, etc.).
5. Revoked by the competent administrative department, etc.

ELIGIBILITY:
Inclusion Criteria:

* 1.1 Aged 14-65 from the outpatients who presented with influenza-like illness (ILI).ILI was defined as a sudden onset of fever (≥ 38°C) with respiratory tract symptoms and at least one of the following symptoms: muscle ache, headache, extreme fatigue or poor activity.

1.2 Confirmed infection by the influenza A or B virus or the new influenza A (H1N1) virus according to virological examination.

1.3 Acute onset within 72 hours. 1.4 Axillary temperature ≥38℃, with at least two of the following symptoms, headache, body discomfort, muscle pain, aversion to cold or cold chills, fatigue; along with either one of the respiratory symptoms from cough, sore throat and nasal symptoms.

1.5 Voluntarily signed informed consents

Exclusion Criteria:

* With one of the following are excluded from the study. 2.1 Aged <14 or >65. 2.2 Chest imaging (X-ray or CT) confirmed bronchitis, pneumonia, pleural effusion, interstitial lesions, etc.

2.3 Routine blood test when screening displayed WBC>10.0x109/L, or NEUT. ≥75%. 2.4 Patients coughing purulent sputum or with suppurative tonsillitis. 2.5 Patients with diabetes or serious underlying disease, such as blood disease, severe COPD (FEV1 / EVC < 70%, FEV1 of expected value < 50%; or respiratory failure or right heart failure), severe hepatic insufficiency (ALT or AST 3 times above normal or higher); severe renal insufficiency (serum creatinine > 2 mg/dL); chronic congestive heart failure (NYHA heart function level Ⅲ- IV), psychiatric diseases.

2.6 Have already taken antiviral drugs (amantadine, rimantadine, zanamivir and oseltamivir phosphate, etc.) or related Chinese medicine or Chinese patent medicine after the onset before the screening. Or patients have taken Choulingdan or Chinese patent medicine with Choulingdan as part of the ingredients within 1 week before the onset.

2.7 Allergic to Choulingdan or its preparations composition, to oseltamivir or its ingredients, and to drug simulation ingredients, or allergic constitution.

2.8 Women in pregnancy or lactation period, women of childbearing age with plan of a pregnancy.

2.9 Patients with immune deficiency, such as malignant tumor, organ or bone marrow transplantation and AIDS, or taking immunosuppressant in 3 months.

2.10 With dubious or confirmed alcohol and drug abuse history. 2.11 Patients that have been in a similar drug clinical study in 3 months. 2.12 Suffered from acute respiratory infection, otitis media or sinusitis 2 weeks before.

2.13 Having vaccination of a seasonal or new influenza A (H1N1) vaccine 6 mouths before.

2.14 Other reasons that researchers think not fitting to participate in the study.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The time needed for alleviation of all influenza symptoms | Up to 30 days
  fever,nasal obstruction, running nose, sore throat, cough, myalgia, fatigue, headache, aversion to cold and sweating

SECONDARY OUTCOMES:
The time of body temperature drop to normal | Up to 30 days
  The time needed for defervescence from the first dose of study medication to the time when body temperature drop to normal (body temperature drop to 37.4℃ or below and is sustained for ≥24 hours)
Total Area Under Curve scores of influenza-like symptoms other than fever | Up to 30 days
  aversion to cold, nasal congestion, muscle aches, sore throat, runny nose, fatigue, headache, cough, sweating
Time to return to normal states of health and activity | Up to 30 days
  Time to return to normal states of health and activity. Return to normal status was defined as the time (in hours) from study drug initiation to the first 24-hour period in which participants returned to their normal state (work or school) and remained so for 24 hours.
Duration of viral shedding (days) | Up to 30 days
  defined as the time from the beginning of study medication to the first time the viral nucleic acid test was negative (negative for both virus culture and PCR, and continuing negative in subsequent virus detection).
The frequency of symptomatic treatment | Up to 30 days
  The frequency of symptomatic treatment
The incidence of influenza complications | Up to 30 days
  The incidence of influenza complications

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Wang, PhD, Study Chair — The 1st Affiliated Hospital of Guangzhou Medical University; Hongixa Ma, PhD, Principal Investigator — The 1st Affiliated Hospital of Guangzhou Medical University

REFERENCES:
- [Derived] He J, Li Z, Huang W, Guan W, Ma H, Yang ZF, Wang X. Efficacy and safety of Chou-Ling-Dan granules in the treatment of seasonal influenza via combining Western and traditional Chinese medicine: protocol for a multicentre, randomised controlled clinical trial. BMJ Open. 2019 Apr 2;9(4):e024800. doi: 10.1136/bmjopen-2018-024800. PMID 30944133